CLINICAL TRIAL: NCT02591342
Title: Comparison of a Cemented, Polished Tapered Stem and an Anatomic Stem for Femoral Neck Fracture
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SM_IV
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hip Fracture; Femoral Neck Fracture; Periprosthetic Femoral Fracture
Keywords: femoral neck fracture; hip arthroplasty; complication; periprosthetic femoral fracture
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CPT stem: Patients treated with a polished, tapered femoral stem as a hip arthroplasty for a displaced femoral neck fracture
- SP2 stem: Patients treated with a anatomic femoral stem as a hip arthroplasty for a displaced femoral neck fracture

SUMMARY:
Postoperative periprosthetic femoral fracture after hip arthroplasty is associated with considerable morbidity and mortality. Recent cohort studies have demonstrated a high incidence of PPF in elderly patients treated with two commonly used polished, tapered, collarless stems in elderly patients. The aim of this study was to compare the rate and characteristics of PPF in a consecutive cohort of patients treated either the polished tapered CTP stem or the matte anatomic SP2 stem in an elderly population above 80 years of age with femoral neck fracture.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Treated with a primary hip arthroplasty

Exclusion Criteria:

* Secondary arthroplasty due to sequel after femoral fracture

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We included all patients above the age of 80 years old, operated between September 2009 and April 2015 with a primary hip arthroplasty for an acute displaced femoral neck fractures. Patients were treated either with the cemented CPT or SP2 stems.
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2009-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of periprosthetic femoral fracture | 2 years

SECONDARY OUTCOMES:
Type of periprosthetic femoral fracture | 2 years
Type of complications after surgery for periprosthetic femoral fracture | 2 years
Mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mukka, M.D, PhD, Principal Investigator — Umeå University

REFERENCES:
- [Background] Broden C, Mukka S, Muren O, Eisler T, Boden H, Stark A, Skoldenberg O. High risk of early periprosthetic fractures after primary hip arthroplasty in elderly patients using a cemented, tapered, polished stem. Acta Orthop. 2015 Apr;86(2):169-74. doi: 10.3109/17453674.2014.971388. Epub 2014 Oct 3. PMID 25280133
- [Background] Inngul C, Enocson A. Postoperative periprosthetic fractures in patients with an Exeter stem due to a femoral neck fracture: cumulative incidence and surgical outcome. Int Orthop. 2015 Sep;39(9):1683-8. doi: 10.1007/s00264-014-2570-0. Epub 2014 Oct 24. PMID 25341951
- [Background] Thien TM, Chatziagorou G, Garellick G, Furnes O, Havelin LI, Makela K, Overgaard S, Pedersen A, Eskelinen A, Pulkkinen P, Karrholm J. Periprosthetic femoral fracture within two years after total hip replacement: analysis of 437,629 operations in the nordic arthroplasty register association database. J Bone Joint Surg Am. 2014 Oct 1;96(19):e167. doi: 10.2106/JBJS.M.00643. PMID 25274795